CLINICAL TRIAL: NCT03321695
Title: An Observational Study of the Safety of Atezolizumab in Patients With Locally Advanced or Metastatic Non Small Cell Lung Cancer in Argentina
Brief Title: A Study of the Safety of Atezolizumab in Participants With Locally Advanced or Metastatic Non Small Cell Lung Cancer in Argentina
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML39852
Record Dates: First submitted 2017-10-20; First posted 2017-10-26 (Actual); Last update posted 2023-03-13 (Actual); Status verified 2023-03

CONDITIONS: Carcinoma, Non-small-cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a study of the safety and effectiveness of atezolizumab in participants with metastatic non-small cell lung cancer (NSCLC) who have disease progression during or following platinum-containing chemotherapy. Participants also will have progressed on an appropriate approved targeted therapy if their tumor has epidermal growth factor receptor (EGFR) or anaplastic lymphoma kinase (ALK) gene abnormalities treated in common clinical practice settings in Argentina.

ELIGIBILITY:
Inclusion Criteria:

* Signed an informed consent form submitted to the Administración Nacional de Medicamentos Alimentos y Tecnología Médica (ANMAT)
* Locally advanced or metastatic (Stage IIIB, Stage IV, or recurrent) non-small cell lung cancer (NSCLC)
* Have received at least one dose of atezolizumab as per local label and clinical practice

Exclusion Criteria:

* Contraindicated atezolizumab therapy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will include participants with locally advanced or metastatic (Stage IIIB, Stage IV, or recurrent) non-small cell lung cancer (NSCLC) who have received the indication for treatment with atezolizumab, as per local label (disease progression during or following treatment with a prior platinum-containing regimen for locally advanced, unresectable/inoperable or metastatic NSCLC or disease recurrence after treatment with a platinum-based adjuvant/neoadjuvant regimen, and have progressed on an appropriate approved targeted therapy if their tumor has EGFR or ALK gene abnormalities) and who have no contraindication to atezolizumab therapy.
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2017-12-27 (Actual); Primary Completion 2019-03-02 (Actual); Study Completion 2019-03-02 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants With Adverse Events | Up to approximately 2 years

SECONDARY OUTCOMES:
Overall Survival (OS) | Up to approximately 2 years
Percentage of Participants With a Confirmed Objective Response (ORR) of Complete Response (CR) or Partial Response (PR) | Up to approximately 2 years
Duration of Response (DOR) | Up to approximately 2 years
Progression-Free Survival (PFS) | Up to approximately 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Productos Roche S.A. Quimica e Industrial, División Farmacéutica, Buenos Aires, Argentina